CLINICAL TRIAL: NCT00323739
Title: Phase II Trial of Bevacizumab(Avastin) and RAD001(Everolimus)in the Treatment of Patients With Advanced Clear Cell Renal Carcinoma
Brief Title: Bevacizumab (Avastin) and RAD001(Everolimus)in the Treatment of Advanced Clear Cell Renal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 32
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Kidney Cancer
Keywords: kidney cancer; bevacizumab
MeSH Terms: conditions — Kidney Neoplasms | interventions — Bevacizumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab and RAD001 (Experimental): Bevacizumab 10mg/kg, IV infusion, every 2 weeks RAD001 10 mg by mouth daily
  Interventions: Drug: bevacizumab; Drug: RAD001

INTERVENTIONS:
Drug: bevacizumab — Bevacizumab 10mg/kg, IV infusion, every 2 weeks
  Other Names: Avastin
Drug: RAD001 — RAD001 10 mg by mouth daily
  Other Names: Everolimus

SUMMARY:
This phase II trial will evaluate the combination of bevacizumab + RAD001 in patients with metastatic renal cell carcinoma. In this trial the investigators will evaluate this combination in patients previously untreated with any anti-angiogenesis agent and patients who have previously received one prior regimen containing an anti-angiogenesis agent.

DETAILED DESCRIPTION:
All eligible patients will receive:

* Bevacizumab 10mg/kg, IV infusion, every 2 weeks
* RAD001 10 mg by mouth daily

All patients will be evaluated for response after completing two courses (8 weeks) of treatment. Patients with objective tumor response or stable disease will continue treatment with bevacizumab adn RAD001 on the same schedule. Treatment will continue until disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic or unresectable locally recurrent clear cell renal carcinoma.
* In patients with mixed histologies, the clear cell component must comprise ≥ 75% of the cancer
* Previous nephrectomy is required with the following exceptions:
* Primary tumor < 5cm
* Extensive liver ( > 30% of liver parenchyma)or
* Multiple (> 5) bone metastases, making nephrectomy a clinically contraindicated procedure
* Patients may have had a maximum of 1 previous systemic regimen for metastatic disease
* Patients may not have received previous bevacizumab. However, patients who have received other agents with anti-angiogenic activity (eg. sorafenib, SU11248, AG-013736, PTK787, thalidomide) as part of first-line treatment are eligible
* Patients may not have received previous treatment with m-TOR inhibitors.
* ECOG performance status 0 or 1
* Measurable disease
* Adequate liver, kidney and bone marrow function
* No previous systemic treatment or radiation therapy for at least 2 weeks prior to study entry
* Patients must be able to understand the nature of this study and give written informed consent

Exclusion Criteria:

* Age < 18 years
* Treatment with > 1 previous systemic regimen for metastatic renal carcinoma
* History of acute myocardial infarction within 6 months
* Clinically significant cardiovascular disease
* History of stroke within 6 months
* Patients with active brain metastases
* Patients with meningeal metastases
* Women who are pregnant or lactating
* Patients who have been treated within 5 years for other invasive cancers
* Patients with history or evidence by physical examination of CNS disease
* Patients with clinical history of hemoptysis or hematemesis
* Patients with history of deep vein thrombosis or thromboembolic disease requiring full dose anticoagulation
* Patients with major surgical procedures, open biopsies, or significant traumatic injuries within 28 days or anticipated need for major surgical procedure during the course of the study
* Patients with peg-tubes or G-tubes
* Patients are ineligible if a fine needle aspiration biopsy has been performed within seven days
* Patients with proteinuria
* Patients with any non-healing wound, ulcer, or long-bone fracture
* Patients with any history of a bleeding diathesis or coagulopathy
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months
* Patients who have received any other experimental drug within 28 days of starting treatment
* History of any other severe and/or uncontrolled medical disease
* History of HIV infection
* Chronic treatment with steroids or other immunosuppressive agents
* Patients with impaired GI function that compromises the ability to swallow or absorb RAD001
* Patients who are unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-05; Primary Completion 2008-11 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (12):
- United States (12):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Gainsville Hematology Oncology Associates, Gainesville, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Wellstar Cancer Research, Marietta, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Methodist Cancer Center, Omaha, Nebraska
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Burris HA 3rd, Waterhouse D, Clark BL, Whorf R. Phase II trial of bevacizumab and everolimus in patients with advanced renal cell carcinoma. J Clin Oncol. 2010 May 1;28(13):2131-6. doi: 10.1200/JCO.2009.26.3152. Epub 2010 Apr 5. PMID 20368560

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-four patients with advanced kidney cancer were assessed for participation at multiple US clinics between August 2006 and November 2008.
Pre-assignment Details: Four patients did not meet eligibility criteria and were not treated.
Groups:
- Bevacizumab and Everolimus: Patients received 10mg/kg of bevacizumab by IV infusion on day 1 and day 15 of each 28-day treatment cycle. Patients took 1 10mg tablet of everolimus every day for 28 days. Treatment continued until evidence of their disease worsening was found or until the side effects of treatment became intolerable to the patient. The treating physician could also stop treatment if the patient's safety was felt to be at risk.
Period: Overall Study
Arm/Group | Bevacizumab and Everolimus
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Everolimus
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 60
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Everolimus
Number analyzed (Participants) | 80
Months | 8.1 [6.3 to 10.8]

2. Secondary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab and Everolimus
Number analyzed (Participants) | 80
Months | 18.5 [14.52 to NA] — Patients remained on treatment at the time statistical analyses were conducted.

ADVERSE EVENTS:
Arm/Group | Bevacizumab + Everolimus
Serious Adverse Events (participants affected / at risk) | 25/80
Other Adverse Events (participants affected / at risk) | 62/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Everolimus (N=80)
Ventricular arrhythmia - left ventricular dysfunction (Cardiac disorders) | 1 (1)
Mood alteration - depression (Psychiatric disorders) | 1 (1)
Thrombus/thrombosis/embolism - lung (Vascular disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 2 (2)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2)
Inflammation - small bowel (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Fracture - right hip (Injury, poisoning and procedural complications) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Obstruction - small bowel (Gastrointestinal disorders) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Obstruction - bowel (Gastrointestinal disorders) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Infection - pneumonia (Infections and infestations) | 2 (2)
Abcess - lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Pneumonitis (non-infectious) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Infection, not otherwise specified (Infections and infestations) | 1 (1)
Parapneumonic effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pain - abdomen (General disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Injury - compression of right mainstem bronchus (Injury, poisoning and procedural complications) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection - urosepsis (Infections and infestations) | 1 (1)
Perforation - rectum (Gastrointestinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Hemmorhage - rectum (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Weakness (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Everolimus (N=80)
Alk Phosphate (Metabolism and nutrition disorders) | 17 (32)
Anorexia (Gastrointestinal disorders) | 27 (94)
AST,SGOT (Metabolism and nutrition disorders) | 11 (24)
Asthenia (General disorders) | 6 (11)
Chills (General disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 19 (47)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (54)
Creatinine (Metabolism and nutrition disorders) | 26 (166)
Dehydration (Gastrointestinal disorders) | 13 (15)
Diarrhea (Gastrointestinal disorders) | 35 (98)
Dizziness (Nervous system disorders) | 8 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (125)
Edema (Blood and lymphatic system disorders) | 18 (58)
Edema (limb) (Blood and lymphatic system disorders) | 14 (45)
Fatigue (General disorders) | 62 (359)
Fever (General disorders) | 12 (22)
Hematuria (Renal and urinary disorders) | 4 (41)
Hemoglobin (Blood and lymphatic system disorders) | 51 (444)
Hemorrhage (nose) (Vascular disorders) | 25 (107)
Hemorrhoids (Gastrointestinal disorders) | 6 (16)
Hypercalcemia (Metabolism and nutrition disorders) | 7 (10)
Hypercholesterolemia (Metabolism and nutrition disorders) | 33 (162)
Hyperglycemia (Metabolism and nutrition disorders) | 24 (76)
Hyperlipidemia (Metabolism and nutrition disorders) | 4 (8)
Hypertension (Cardiac disorders) | 34 (143)
Hypoalubminemia (Metabolism and nutrition disorders) | 6 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (21)
Hypokakalemia (Metabolism and nutrition disorders) | 7 (14)
Hyponatremia (Metabolism and nutrition disorders) | 6 (22)
Infection (NOS) (Infections and infestations) | 5 (7)
Infection (sinus) (Respiratory, thoracic and mediastinal disorders) | 5 (24)
Infection (URI) (Respiratory, thoracic and mediastinal disorders) | 9 (15)
Infection (UTI) (Renal and urinary disorders) | 9 (12)
Leukocytes (WBC) (Blood and lymphatic system disorders) | 21 (142)
Mental Status Change (Nervous system disorders) | 4 (5)
Mood alteration (anxiety) (Nervous system disorders) | 7 (27)
Mood alteration (depression) (Nervous system disorders) | 12 (81)
Mucositis (Gastrointestinal disorders) | 35 (102)
Nail Changes (Skin and subcutaneous tissue disorders) | 4 (12)
Nausea (Gastrointestinal disorders) | 33 (92)
Neuropathy (Nervous system disorders) | 4 (9)
Neuropathy (sensory) (Nervous system disorders) | 6 (14)
Neutrophils (ANC) (Blood and lymphatic system disorders) | 13 (55)
Pain (abdominal) (Gastrointestinal disorders) | 8 (14)
Pain (back) (Musculoskeletal and connective tissue disorders) | 12 (64)
Pain (bone) (Musculoskeletal and connective tissue disorders) | 6 (10)
Pain (chest) (Cardiac disorders) | 15 (38)
Pain (headache) (Nervous system disorders) | 25 (82)
Pain (jaw) (Musculoskeletal and connective tissue disorders) | 4 (7)
Pain (joint) (Musculoskeletal and connective tissue disorders) | 10 (60)
Pain (limb) (Musculoskeletal and connective tissue disorders) | 21 (107)
Pain (myalgia) (Musculoskeletal and connective tissue disorders) | 11 (34)
Pain (neck) (Musculoskeletal and connective tissue disorders) | 7 (19)
Pain (NOS) (General disorders) | 16 (41)
Pain (oral) (Gastrointestinal disorders) | 4 (4)
Pain (throat) (Gastrointestinal disorders) | 9 (19)
Phosphorous (Metabolism and nutrition disorders) | 6 (8)
Platelets (Blood and lymphatic system disorders) | 32 (225)
Proteinuria (Metabolism and nutrition disorders) | 36 (243)
Pruritis (Skin and subcutaneous tissue disorders) | 16 (55)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 37 (122)
Reflux (Gastrointestinal disorders) | 6 (81)
Skin (erythema) (Skin and subcutaneous tissue disorders) | 10 (51)
Skin (lesion) (Skin and subcutaneous tissue disorders) | 5 (20)
Sore (mouth) (Gastrointestinal disorders) | 4 (6)
Stomatitis (Gastrointestinal disorders) | 14 (26)
Tachycardia (Cardiac disorders) | 4 (9)
Taste Alteration (Gastrointestinal disorders) | 12 (35)
Triglycerides (Metabolism and nutrition disorders) | 32 (190)
Uric acid (Metabolism and nutrition disorders) | 9 (32)
Voice change (Respiratory, thoracic and mediastinal disorders) | 8 (41)
Vomiting (Gastrointestinal disorders) | 14 (37)
Weakness (General disorders) | 15 (32)
Weight Loss (General disorders) | 13 (41)
Infection (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Insomnia (General disorders) | 14 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.